CLINICAL TRIAL: NCT02422550
Title: Development and Evaluation of Imaging Acquisition and Analysis Methods for Optimization of MRI and/or CT in Radiation Oncology Simulation, Treatment Planning, and Response Assessment
Brief Title: Imaging Acquisition and Analysis Methods for Optimization of MRI Radiation Oncology Simulation and Response Assessment
Status: Recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 15-073
Record Dates: First submitted 2015-04-14; First posted 2015-04-21 (Estimated); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Radiation Therapy
Keywords: MRI; 15-073; participants undergoing radiation therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- participants undergoing radiation therapy & normal volunteers: Protocol participation will consist of one or more research MRI or CT exams not to exceed 45 minutes.
  Interventions: Device: MRI or CT

INTERVENTIONS:
Device: MRI or CT — Participants enrolled on this protocol may undergo multiple MRI or CT examinations periodically over the course of their treatment and follow-up if they are participating in a development project related to tumor response assessment. Volunteers enrolled on this protocol may undergo multiple MRI examinations periodically for studies of reproducibility.

SUMMARY:
Magnetic resonance imaging (MRI) is currently one of the standard diagnostic imaging methods used to diagnose tumor stage before treatment in the Radiation Oncology Department. It is also used to check responses to radiation after treatment. However, MRI isn't traditionally used in planning for radiation treatment or in checking treated tumor and tissue changes during radiation treatment. The goal is to find out the possible benefits of MRI imaging techniques in these settings of radiation treatment. The research aims are to study the possibility of using devices with new abilities such as the MR-Linac. The MR-Linac combines a radiation treatment machine with a diagnostic MRI scanner. This device will improve the quality of MRI-guided radiation treatment. The MR-Linac has functions that are currently not available in other combined imaging and radiation delivery devices. The MR-Linac does not provide additional imaging capabilities that are not currently available in other imaging devices.

Participating in this study would NOT change the current treatment plans, this will allow the investigators to use the MRI methods in research and future patient care.

DETAILED DESCRIPTION:
The purpose of this protocol is to demonstrate proof of concept and feasibility of new MRI or CT hardware, pulse sequences and data analysis software to plan and adapt radiotherapy treatment and to assess tumor response to radiotherapy (only FDA approved hardware are allowed in this study). Efforts to develop, modify and evaluate new or existing MR or CT imaging techniques must be a continuous practice with the goal of enhancing the use of MRI or CT during radiation therapy. The investigators therefore anticipate an ongoing need for such a protocol and believe the ability to perform such studies is critical to the translation of new imaging technologies from concept to routine clinical use. Under this protocol, modifications to the following items may be tested: pulse sequence programs, radiofrequency coils, reconstruction and processing software, other MR or CT system hardware and analysis software. A brief description of each of these items is described below. The potential risks associated with modifying each of these items, and the measures that will be taken to minimize these risks are described in subsequent sections.

ELIGIBILITY:
Inclusion Criteria:

* Men and women age 18 or older

Exclusion Criteria:

* Anyone who would be normally excluded from undergoing an MRI examination as per Memorial Hospital for Cancer and Allied Diseases Screening Questionnaire
* Participants/volunteers with a pacemaker, aneurysm clip or any other condition that would warrant avoidance of a strong magnetic field
* Female participants/volunteers who are pregnant or nursing
* Participants/Volunteers who are unable to comply or complete the MRI exam due to claustrophobia or high levels of anxiety
* Participants/Volunteers from the vulnerable population, as defined by 45 CFR 46.
* Participants at higher risk due to age, frailty, or the emergent nature of their condition.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population will be participants undergoing radiation therapy in the Department of Radiation Oncology, optional normal volunteers, or a combination thereof.
Sampling Method: Non-Probability Sample
Enrollment: 837 (Estimated)
Dates: Start 2015-04-09 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
evaluate the feasibility of new MRI or CT applications | 5 years
  MRI or CT acquisition and analysis methods for radiotherapy planning or tumor response assessment during radiotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Lee, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering Basking Ridge (Consent only), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Consent only), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Consent only ), Montvale, New Jersey
  - Memorial Sloan Kettering Commack (Consent Only), Commack, New York
  - Memorial Sloan Kettering Westchester (Consent only), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Consent only), Uniondale, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://one.mskcc.org/sites/pub/Pages/default.aspx